CLINICAL TRIAL: NCT05651750
Title: Medical vs Surgical Treatment Decision in Pediatric Obstructive Sleep Apnea Using Sleep Questionnaire
Brief Title: Medical vs Surgical Treatment in OSA Among Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Assaf-HarofehMC
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2021-12

CONDITIONS: To Evaluate PSQ as Clinical Tool in the Decision Between Medical and Surgical Treatment for Adenotonsillar Hypertrophy; To Determine Clinical Response to Montelukast or Nasal Steroids Based on PSQ Results
MeSH Terms: interventions — montelukast; fluticasone furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Montelukast tab (Experimental)
  Interventions: Drug: Montelukast
- Fluticasone nasal spray (Experimental)
  Interventions: Drug: Fluticasone Furoate

INTERVENTIONS:
Drug: Montelukast — receiving 2 months treatment with Montelukast once a day
  Other Names: Singulair
  Arms: Montelukast tab
Drug: Fluticasone Furoate — receiving 2 months treatment with Fluticasone Furoate nasal spray once a day
  Other Names: Avamys
  Arms: Fluticasone nasal spray

SUMMARY:
Adeno-tonsillar hypertrophy causing OSA are treated surgically however, over the last years it has been shown that montelukast or nasal steroidal spray can significantly improve symptoms, adenoid size, and polysomnographic results in pediatric non-severe OSA, excluding the need for surgery. A literature review from 2016 suggested that by using anti-leukotrienes as anti-inflammatory appears to be beneficial in children with a non-severe OSA and can be offered to parents as a treatment option before, or instead of surgery. In addition, nasal steroidal spray may be considered useful in decreasing adenoid pad size and the severity of symptoms related to adenoidal hypertrophy [9]. Despite emerging evidence that both montelukast and nasal steroids are effective in the treatment of pediatric SDB, further evidence is still required. . adeno-tonsillar hypertrophy causing OSA are treated surgically however, over the last years it has been shown that montelukast or nasal steroidal spray can significantly improve symptoms, adenoid size, and polysomnographic results in pediatric non-severe OSA, excluding the need for surgery. A literature review from 2016 suggested that by using anti-leukotrienes as anti-inflammatory appears to be beneficial in children with a non-severe OSA and can be offered to parents as a treatment option before, or instead of surgery. In addition, nasal steroidal spray may be considered useful in decreasing adenoid pad size and the severity of symptoms related to adenoidal hypertrophy. Despite emerging evidence that both montelukast and nasal steroids are effective in the treatment of pediatric SDB, further evidence is still required.

ELIGIBILITY:
Inclusion Criteria:

* children between 2-16 years of age referred to the pediatric otolaryngology outpatient clinic due to OSA and have not undergone previous adeno-tonsillar procedure

Exclusion Criteria:

* children with severe OSA who need an urgent surgery and cannot be postponed, children with nasal polyposis, craniofacial malformations (e.g. cleft lip and palate), and genetic diseases (e.g. Down syndrome).

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate PSQ as clinical tool in the decision between medical vs surgical treatment for adeno-tonsillar hypertrophy | 1 year

SECONDARY OUTCOMES:
To determine clinical response to montelukast or nasal steroids based on PSQ results | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Be’er Ya‘aqov, Israel